CLINICAL TRIAL: NCT07321106
Title: A Phase 1, First-in-human (FIH), Dose-Escalation and Dose-Optimization Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Anti-tumor Activity of CBI-1214 T Cell Engager in Participants With Advanced or Metastatic Microsatellite Stable (MSS)/Microsatellite Instability Low (MSI-L) Colorectal Cancer
Brief Title: A Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Anti-tumor Activity of CBI-1214 T Cell Engager in Participants With Advanced or Metastatic MSS/MSI-L Colorectal Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cartography Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CBI-1214-001
Record Dates: First submitted 2025-12-15; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Cancer; Colorectal Cancer (CRC); Colorectal (Colon or Rectal) Cancer; CRC; Metastatic Colon Cancer; Colon Cancer; Advanced Colorectal Cancer
Keywords: Oncology; Solid Tumor; Phase 1; First-in-Human; Dose Escalation; Open-Label; T-Cell Engager; TCE
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose escalation and optimization trial of CBI-1214 (Experimental): Participants will be assigned sequentially to escalating doses of CBI-1214. Once dose escalation is completed, a recommended expansion dose will be proposed for the dose-expansion stage of the trial.
  Interventions: Biological: CBI-1214

INTERVENTIONS:
Biological: CBI-1214 — CBI-1214 is a bispecific T cell engager that binds to LY6G6D and CD3. It is designed to link the patients T cells to cancer cells and to mediate tumor cell killing. LY6G6D is an emerging target specifically expressed on malignant colorectal cancer cells.

SUMMARY:
This study will investigate the safety, tolerability, pharmacokinetics, and anti-tumor activity of CBI-1214 in participants with advanced or metastatic Microsatellite Stable (MSS)/Microsatellite Instability Low (MSI-L) Colorectal Cancer

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Participant with MSS/MSI-L CRC, who has exhausted at least one prior line of standard systemic therapy for their current malignancy.
* Participant with genomic aberrations, including but not limited to BRAFV600E mutations and HER2 amplifications, for which FDA-approved targeted therapies are available, must:

  * Have received prior treatment with applicable FDA-approved targeted therapies AND
  * Either have experienced disease progression, be refractory, or be intolerant to directed molecular therapy.
* Participant able to provide archival tissue sample or fresh biopsy tissue sample

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Participant whose CRC tumor tissues have been identified as dMMR or MSI-H
* Known history of solid organ or tissue transplant; history of interstitial lung disease or non-infectious pneumonitis.
* Untreated central nervous system (CNS) metastatic disease.
* Active autoimmune disease that has required systemic treatment within the past 2 years (participants with hormone replacement therapy for adequately controlled endocrinopathy are allowed in the study).
* History of recent infection (within 4 weeks of C1D1) considered to be caused by one of the pathogens: HSV1, HSV2, VZV, EBV, CMV, measles, Influenza A, Zika virus, Chikungunya virus, mycoplasma pneumonia, Campylobacter jejuni, or enterovirus D68.
* Known seropositive for human immunodeficiency virus, hepatitis B surface antigen, or antibody to hepatitis C virus with confirmatory testing and requiring anti-viral therapy.
* History of Steven's Johnson's syndrome or toxic epidermal necrolysis syndrome.
* Significant medical comorbidities, including uncontrolled hypertension (diastolic blood pressure >115 mm Hg), unstable angina, congestive heart failure (greater than New York Heart Association class II), severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia, poorly controlled diabetes, severe chronic pulmonary disease, coronary angioplasty, or myocardial infarction within 6 months prior to screening, or uncontrolled atrial or ventricular cardiac arrhythmias.
* Congenital long QT syndrome or a corrected QT interval (QTc) ≥480 ms at screening (unless secondary to pacemaker or bundle branch block).
* Active second primary malignancy within 3 years of Screening other than non-melanoma skin cancers, nonmetastatic prostate cancer, in situ cervical cancer, or ductal or lobular carcinoma in situ of the breast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-04 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of CBI-1214 at increasing dose levels and optimized dose levels in participants with advanced or metastatic MSS/MSI-L CRC | Approximately 48 months
  Incidence and severity of TEAEs, TRAEs, and TESAEs; changes in vital signs, physical examinations, and clinical laboratory parameters per NCI-CTCAE v5.0.
To determine the MTD and/or OBD and select the recommended dose(s) of CBI-1214 for dose optimization | Approximately 48 months
  Incidence of DLTs observed during the first treatment cycle

SECONDARY OUTCOMES:
To characterize the Serum Concentration of CBI-1214. | Approximately 48 months
  Serum concentration of CBI-1214 at specified timepoints following a single infusion as well as following repeat infusions.
Overall Response Rate (ORR) | Approximately 48 months
  ORR is defined as the proportion of patients with a complete response (CR) or partial response (PR) as determined by the investigator according to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1)
Duration of Response (DOR) | Approximately 48 months
  Duration of response (DOR), defined as the time from the first occurrence of a documented objective response to disease progression or death from any cause (whichever occurs first), as determined by the investigator according to RECIST v1.1
Progression Free Survival (PFS) | Approximately 48 months
  The time from the date of first dose of study treatment to the first documentation of disease progression as determined by RECIST version 1.1, or death from any cause, whichever occurs first.
Time to Response (TTR) | Approximately 48 months
  The time from the date of first dose of study treatment to the first documented evidence of objective tumor response (Complete Response [CR] or Partial Response [PR]) as assessed per RECIST version 1.1.
Clinical Benefit Rate (CBR) | Approximately 48 months
  The proportion of subjects who achieve Complete Response (CR), Partial Response (PR), or Stable Disease (SD) lasting for a minimum prespecified duration (e.g., ≥12 or ≥16 weeks) as determined by RECIST version 1.1.
Overall Survival (OS) | Approximately 48 months
  The time from the date of first dose of study treatment to death from any cause.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - NEXT Oncology, San Antonio, Texas
  - NEXT Oncology, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No